CLINICAL TRIAL: NCT00160459
Title: A Phase 2, Randomized, Double-Blind, Parallel Group Study to Evaluate the Safety and Efficacy of Asoprisnil (J867) in Patients With Uterine Leiomyomata.
Brief Title: A Study to Evaluate the Safety and Effectiveness of Asoprisnil in the Treatment of Uterine Fibroids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Cynthia Mattia-Goldberg, Abbott
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M99-144
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Leiomyoma
Keywords: Fibroid Uterus; Leiomyoma; Uterine Fibroids; asoprisnil
MeSH Terms: conditions — Leiomyoma | interventions — asoprisnil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Asoprisnil
- 2 (Experimental)
  Interventions: Drug: Asoprisnil
- 3 (Experimental)
  Interventions: Drug: Asoprisnil
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Asoprisnil — 5 mg Tablet, oral Daily for 12 weeks
  Arms: 1
Drug: Asoprisnil — 10 mg Tablet, oral Daily for 12 weeks
  Arms: 2
Drug: Asoprisnil — 25 mg Tablet, oral Daily for 12 weeks
  Arms: 3
Drug: Placebo — Tablet, oral Daily for 12 weeks
  Arms: 4

SUMMARY:
This study was designed to determine the safety and effectiveness of 3 asoprisnil doses compared to placebo, taken for 12 weeks by women with uterine fibroids.

DETAILED DESCRIPTION:
No medical therapy is currently available for the long-term treatment of uterine fibroids. The objective of this study is to determine the safety and efficacy of asoprisnil 5 mg, 10 mg and 25 mg, compared to placebo, taken daily for 12 weeks by women with one or more uterine fibroids, confirmed by ultrasound. Upon completion, subjects at participating sites will be allowed to enter an open-label extension study

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 49 years of age
* Diagnosis of either 1 or more uterine fibroids
* History of regular menstrual cycles of 21 to 35 days in length.

Exclusion Criteria:

* Any abnormal lab result the study-doctor considers significant
* History of severe reaction to or current use of hormone therapy
* History of osteoporosis or other bone disease
* History of uterine artery embolization, cryomyolysis, or electrical myolysis
* Subject currently breast feeding
* Hemoglobin < 8 g/dL at baseline

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2000-05; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in uterine volume and volume of the largest fibroid. | Treatment weeks 4, 8, 12 and Post-treatment months 3 and 6.
Duration of amenorrhea | Day 1 to 1st post treatment menses

SECONDARY OUTCOMES:
Change from baseline in uterine size in gestational weeks. | Treatment weeks 4, 8, 12 and Post-treatment months 3 and 6
Number of Subjects in each treatment group achieving> or = to 20% reduction in uterine volume. | Week 12 and final visit
Percentage of days with bleeding. | Day 1 through end of 1st post-treatment menses
Changes in hematologic and iron parameters. | Baseline to each visit
Uterine fibroid symptom improvement. | Baseline to each visit
Response to Global Efficacy Question regarding improvement in fibroid symptoms. | Week 12 and Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Abbott

REFERENCES:
- [Result] Chwalisz K, Larsen L, Mattia-Goldberg C, Edmonds A, Elger W, Winkel CA. A randomized, controlled trial of asoprisnil, a novel selective progesterone receptor modulator, in women with uterine leiomyomata. Fertil Steril. 2007 Jun;87(6):1399-412. doi: 10.1016/j.fertnstert.2006.11.094. Epub 2007 Feb 20. PMID 17307170